CLINICAL TRIAL: NCT00728429
Title: CCCWFU 99108 - Effect of Exercise Training in Patients Receiving Anthracycline Drugs - A Pilot Study
Brief Title: Aerobic Exercise in Patients Receiving Chemotherapy for Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000601334; CCCWFU-99108; CCCWFU-IRB-IRB00006209
Record Dates: First submitted 2008-08-02; First posted 2008-08-05 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Toxicity; Chemotherapeutic Agent Toxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cardiac toxicity; chemotherapeutic agent toxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): normal anthracycline therapy
- exercise program (Experimental)
  Interventions: Behavioral: exercise intervention

INTERVENTIONS:
Behavioral: exercise intervention — 24 week program of exercise
  Arms: exercise program

SUMMARY:
RATIONALE: Aerobic exercise may help prevent side effects caused by chemotherapy and help improve heart health.

PURPOSE: This randomized clinical trial is studying the side effects of aerobic exercise and to see how well it works in patients receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if patients with cancer can exercise safely and routinely, under supervision, while receiving anthracycline chemotherapy.
* To determine the magnitude of the change in the peak ventilatory oxygen uptake (VO2) before and after completion of anthracycline chemotherapy with concurrent exercise versus without exercise in patients with cancer.

OUTLINE: Patients are randomized to 1 of 2 intervention arms.

* Arm I (exercise): Patients undergo supervised aerobic exercise (walk or bicycle) 3 days a week concurrently with standard anthracycline-based chemotherapy for approximately 18-24 weeks.
* Arm II (non-exercise): Patients receive standard anthracycline-based chemotherapy for approximately 18-24 weeks.

Patients undergo peak ventilatory oxygen uptake (VO_2) by exercise bike test with gas exchange analysis at baseline and at 2 weeks after completion of anthracycline-based chemotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with cancer scheduled to receive 4-6 courses of an anthracycline-based chemotherapy

PATIENT CHARACTERISTICS:

* Able to pedal a stationary bicycle
* No severe hypertension (systolic blood pressure > 220 mm Hg or diastolic blood pressure >120 mm Hg)
* No atrial fibrillation with an uncontrolled ventricular response
* No ventricular arrhythmias
* No unstable angina
* No acute myocardial infarction within the past 28 days of enrollment
* No severe valvular heart disease
* No severe (exercise-limiting) peripheral vascular disease
* No severe pulmonary disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients enrolling in the study | day 1
Percentage of patients completing the study | 24 weeks
V02 peak before and after chemotherapy | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Wells, MD, PhD, Principal Investigator — Wake Forest University Health Sciences; Peter H. Brubaker, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States